CLINICAL TRIAL: NCT03017599
Title: Yield Rate for Procurement the Histologic Core With Endoscopic Ultrasound-guided Fine Needle Biopsy With 20-gauge Ultrasound Biopsy Needles for Solid Pancreatic Masses: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2016-0429
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Pancreatic Cancer; Solid Pancreatic and Peripancreatic Lesion
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): EUS-FNB using 20-gauge procore needle
  Interventions: Device: 20-gauge ProCore FNB needle

INTERVENTIONS:
Device: 20-gauge ProCore FNB needle — The investigators will prospectively collect data base including patients who underwent EUS-guided biopsy with the 20-gauge ProCore histology needle for the evaluation of Pancreatic solid mass.
  EUS procedures will be performed under sedation with linear echoendoscopes. Once the lesion will be penetrated, the stylet will be removed, and suction will be applied for 10 to 20 seconds by using a 10-ml syringe while moving the needle to and fro. All samples will processed at the pathology departments for histological analysis with documentation.
  Other Names: 20G Echotip ProCore Fine Needle Biopsy (FNB) device(Echotip ProCore; Cook Endoscopy Inc, Limerick, Ireland)

SUMMARY:
To investigate the technical feasibility and diagnostic yield of new 20-gauge Procore needle for EUS-guided fine needle biopsy in pancreatic solid lesions.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma is the fourth cause of death in the Western world. Surgery remains the only treatment offering an advantage in terms of overall survival (5-year survival range, 15-25%), but unfortunately only 10-20% of patients present resectable disease at the time of diagnosis.

Regarding the diagnosis of pancreatic cancer, proper tool with high diagnostic yield is very important. The investigators investigated the technical feasibility and diagnostic yield of recent-developed new 20-gauge Procore needle for EUS-guided fine needle biopsy in pancreatic solid lesions.

The investigators applied the 20-gauge procore needle for EUS-guided fine needle biopsy in the diagnosis of pancreatic solid mass. A total of 30 patients will be enrolled for the present pilot study.

ELIGIBILITY:
Inclusion Criteria:

* patients who are at least 20 years of age
* patients who require endoscopic ultrasound-guided fine needle aspiration cytology or biopsy because of pancreatic or peripancreatic solid mass.

Exclusion Criteria:

* Cystic pancreatic mass in imaging tests such as CT or MRI or US
* haemodynamically unstable patients
* severe coagulopathy (international normalized ratio [INR] > 1.5 or platelet count < 50,000 cells/cubic millimeter [cmm3])
* patients unable to quit anticoagulant/anti-platelet therapy
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Procurement of the histologic core | 7 days after the procedure
  The sample quality is evaluated as optimal for histological evaluation; the presence of optimal histological core including recognizable structures
Diagnostic accuracy | 7 days after the procedure
  [Standard diagnosis]
  * In operated patients; based on the surgical resection specimen
  * In non-operated patients; based on the conclusions of the diagnostic work-up and confirmed by a compatible clinical disease course

SECONDARY OUTCOMES:
Technical success | 7 days after the procedure
  Technical failure is defined as malfunction of the needle before the investigators reached a diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JH, Stewart J, Ross WA, Anandasabapathy S, Xiao L, Staerkel G. Blinded prospective comparison of the performance of 22-gauge and 25-gauge needles in endoscopic ultrasound-guided fine needle aspiration of the pancreas and peri-pancreatic lesions. Dig Dis Sci. 2009 Oct;54(10):2274-81. doi: 10.1007/s10620-009-0906-1. Epub 2009 Aug 11. PMID 19669880
- [Background] Siddiqui UD, Rossi F, Rosenthal LS, Padda MS, Murali-Dharan V, Aslanian HR. EUS-guided FNA of solid pancreatic masses: a prospective, randomized trial comparing 22-gauge and 25-gauge needles. Gastrointest Endosc. 2009 Dec;70(6):1093-7. doi: 10.1016/j.gie.2009.05.037. Epub 2009 Jul 28. PMID 19640524